CLINICAL TRIAL: NCT04569045
Title: A Randomized, Within-subject Controlled Clinical Study to Evaluate the Safety and Effectiveness of Pain Relief of Modified Sodium Hyaluronate Gel for Injection When Used for the Correction of Moderate or Severe Nasolabial Folds
Brief Title: Evaluate the Safety and Effectiveness of Sodium Hyaluronate When Used for the Correction of Nasolabial Folds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SciVision Biotech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RDCT-CNFL
Record Dates: First submitted 2020-09-23; First posted 2020-09-29 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2021-02

CONDITIONS: Dermal Filler; Hyaluronic Acid; Lidocaine; Nasolabial Fold

STUDY DESIGN:
Intervention Model Description: Subject's two sides of nasolabial folds (NLF) were randomized to receive FACILLE® Light (contains Lidocaine) or FACILLE® (without Lidocaine).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HA + Lidocaine (Experimental): Sodium Hyaluronate with Lidocaine Hydrochloride
  Interventions: Device: HA+Lidocaine
- HA (Active Comparator): Sodium Hyaluronate
  Interventions: Device: HA

INTERVENTIONS:
Device: HA+Lidocaine — 20 mg
  Arms: HA + Lidocaine
Device: HA — 20 mg
  Arms: HA

SUMMARY:
The aim of this study is to evaluate the safety and effectiveness of pain relief of modified sodium hyaluronate gel for injection when used for the correction of moderate or severe nasolabial folds.

DETAILED DESCRIPTION:
One hundred and thirty patients were enrolled and there two sides of nasolabial folds (NLF) were randomized to receive HA with lidocaine or HA. The primary outcome was immediate visual analogue scale (VAS) of pain evaluated after injection for both NLF sides. Secondary outcomes including VAS pain, wrinkle severity rating scale (WSRS), global aesthetic improvement scale (GAIS) and AE were observed at 1, 3, 6, 9, 12 follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years of male or female
* Wrinkle Severity Rating Scale (WSRS) of bilateral nasolabial folds graded 3 or 4 by blinded evaluator (moderate to severe bilateral nasolabial fold), consistent grade of bilateral nasolabial folds, and the grades approved by the physician who perform the treatment
* Agree not to undergo any other under-eye facial surgery (including nose) during the study period

Exclusion Criteria:

* Injection site with infection or other skin diseases present which may affect the evaluation
* With medical history of chromatosis, discoloration, keloid formation, hypertrophic scarring at nasolabial folds
* With permanent implants or planning to receive permanent implants during the study period at the injection sites
* Hyaluronate facial dermal implant injection or other impermanent dermal fillers injection at injection sites within the past 12 months
* With under-eye facial Botox or fat injection within the past 6 months or planning to receive under-eye facial Botox or fat injection during the study period
* With under-eye facial chemical or lasers peeling, non-invasive skin tightening, thermocool within the past 3 months or planning to receive these aesthetic procedures during the study period
* With prescription medication for nasolabial fold treatment, topical corticosteroid, skinirritating topical products or pigmentation products within the past 2 weeks or planning to take these medication or products during the study period
* With systemic immunosuppressive therapy or systemic corticosteroids within the past 2 months or planning to receive these therapies during the study period (subjects who have received inhaled/intranasal corticosteroids could be considered to include.)
* Severe liver or kidney defects (such as the value of ALT or AST over 1.5 folds of upper limit of normal value; the value of creatinine over 1.5 folds of upper limit of normal value)
* With clinical meaningful coagulation disorders, underdoing anticoagulant treatment or within the past 10 days, or taking blood circulation promotion and blood stasis removement medications
* With epilepsy or porphyria
* With congenital or idiopathic methemoglobinemia or glucose-6-phosphate dehydrogenase deficiency
* With the need to take b-blocker during the study period
* With severe atrioventricular block (type 2 second-degree AV block and third-degree AV block)
* With analgesic dependence, analgesics within the past 2 weeks or planning to receive analgesics during the study period
* With orthodontics, tooth extraction, tooth implantation (extraction or implantation of tooth anterior to the second premolar) or planning to receive these procedures during the study
* With history of hypersensitivity or allergy to lidocaine, amide anesthetics, hyaluronic acid or any component of the device; Gram-positive bacterial or Streptococcus proteins; other severe hypersensitivity history unsuitable for participating in the study
* Planning to undergo any surgery which may cause significant body weight change (such as bariatric surgery) or take any medication which may cause significant body weight change
* Pregnant, planning pregnancy or in breastfeeding females
* With syphilis or HIV infection
* Participated in clinical study of other device or drug and have not terminated within the past 30 days -Other circumstances which judged to be unsuitable for participating in the study by the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2020-12-04 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Immediate VAS pain evaluated after injection for both NLF sides | Immediate post-injection
  The VAS scale uses a 100 mm line labelled at '0' with 'no pain' and '100' with 'worst pain'.

SECONDARY OUTCOMES:
VAS pain evaluated 15, 30, 45 and 60 minutes after injection for both NLF sides | 15, 30, 45 and 60 minutes post-injection
  The VAS scale uses a 100 mm line labelled at '0' with 'no pain' and '100' with 'worst pain'.
On-site WSRS evaluated by site blinded-evaluator at 1, 3, 6, 9 and 12 months | 1, 3, 6, 9 and 12 months post-injection
  Evaluators assess the wrinkle severity of nasolabial folds on site or photographically with 5 graded scale,1 to 5 was represented 'absent' to 'extreme'.
GAIS evaluated photographically by independent blinded-evaluator at 1, 3, 6, 9 and 12 months | 1, 3, 6, 9 and 12 months post-injection
  Evaluators and subjects assess the improvement of correction with 5 graded scale,1 to 5 was represented 'exceptional improvement' to 'worsened'.
Adverse events reported from the baseline and during the study period | 1, 3, 6, 9 and 12 months post-injection
  The safety assessment was based on reports of adverse events, defined as any unwanted events whether it was thought to be related to the study drugs or not, were recorded during each follow up and at any time the patient reported an event to the investigator during the study period.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing, Beijing
  - Shanghai, Shanghai